CLINICAL TRIAL: NCT07036913
Title: Effectiveness of Somatocognitive Therapy With TENS and Stretching Exercises on Menstrual Pain and Quality of Life With Dysmenorrhea.A Randomized Controlled Trial.
Brief Title: Effectiveness of ST With TENS and Stretching Exercises on Menstrual Pain and QOL With Dysmenorrhea. RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1002
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- somatocognitive therapy (Experimental)
  Interventions: Diagnostic Test: somatocognitive therapy
- Stretching exercises (Active Comparator)
  Interventions: Combination Product: Stretching exercises

INTERVENTIONS:
Diagnostic Test: somatocognitive therapy — In somatocognitive therapy which includes drawing( three days prior to menustration in first two months and the first day of menustration in third month) and music(in the first 12 hours of menustration)along with TENS(thirty minutes on abdominal region, upon the onset of dysmonarrhea).
  Arms: somatocognitive therapy
Combination Product: Stretching exercises — Stretching exercises of abdominal, lumbar or pelvic region will be performed as a treatment. Frequency:15 minutes;three times per week.
  Arms: Stretching exercises

SUMMARY:
Effectiveness of somatocognitive therapy with TENS and stretching exercises on menstrual pain and quality of life with dysmenorrhea.A randomized controlled trial The objective of this study is to find weather which therapy; somatocognitive therapy along with TENS or stretching exercises is more effective and what are their effects on quality of life in females with dysmonarrhea.

DETAILED DESCRIPTION:
The Study spans the population into two groups. For first group we will give somatocognitive therapy (drawing and music) along with TENS and in second group we will give stretching exercises. In both groups the hotpack will be the common treatment.

The nature of this study will be randomized controlled trial . We will use simple random sampling technique in this study.

For outcomes measurements we will use numerical rating scale and menustral distress questionere .

ELIGIBILITY:
Inclusion Criteria:

* Females who are facing menustral pain during their every menses.
* Females who are facing dysmonarrhea from the at least last three months.
* Females who are willing to take part in the research.

Exclusion Criteria:

* Females with some hormonal problem.
* Females with irregular menustral cycle.
* Females who face menustral pain during some of their menses
* Pregnant females
* Females with recent abdominal/pelvic surgery.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | 6 Month
  A pain screening tool, commonly use to assess pain severity at that moment in time using a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain".
Menstrual distress questionnaire | 6 Months
  The MSQ is a 24-46 item self-report measure which assesses menstrual pain and symptoms .The score on each item ranges from 1 (never) to 5 (always) with a higher composite score indicating more symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore City, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No